CLINICAL TRIAL: NCT03752762
Title: Effect of an Innovative Behavioral Change Strategy and SQ-LNS on Stunting and Obesity in Children Living in Tepic, Mexico
Brief Title: SPOON: Sustained Program for Improving Nutrition - Mexico
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding cancelled
Sponsor: Inter-American Development Bank (Other)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); The PepsiCo Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Inter-AmericanDB Mexico
Record Dates: First submitted 2018-01-08; First posted 2018-11-26 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Exclusive Breastfeeding; Feeding Patterns; Stunting; Obesity, Childhood
Keywords: Stunting; Obesity; Lipid-based Nutrient Supplements (LNS); Latin America; Child nutrition; Feeding practices
MeSH Terms: conditions — Breast Feeding; Feeding Behavior; Growth Disorders; Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will receive standard health care services provided by the Health Secretary
- SPOON behavioral change strategy+SQ-LNS (Experimental): Participants will receive SQ-LNS supplement from 6-24 months and a behavioral change to promote adequate infant and young child feeding practices and the use of SQ-LNS will be delivered to mothers or caregivers. The behavioral change strategy includes individual home-visits and group sessions. SQ-LNS consists of a 20g nutrient supplement package to be consumed daily from 6-24 of age. SQ-LNS formulation does not include sugar.
  Interventions: Dietary Supplement: SQ-LNS; Behavioral: SPOON behavioral change strategy

INTERVENTIONS:
Dietary Supplement: SQ-LNS — SQ-LNS is a peanut-based ready to use home fortification product to improve diet quality in children 6-24 months of age. It includes peanuts and other ingredients such as vegetable fat, powdered milk and several micronutrients. The formulation designed for this study will not include sugar.
  Other Names: Small Quantity Lipid Nutrient Supplements
  Arms: SPOON behavioral change strategy+SQ-LNS
Behavioral: SPOON behavioral change strategy — An innovative behavioral change strategy designed using ethnographic and marketing methods to promote adequate infant and young child feeding practices and the use of SQ-LNS. The strategy will be delivered to mothers or caregivers through individual home-visits and group sessions.
  Arms: SPOON behavioral change strategy+SQ-LNS

SUMMARY:
The primary goal of this study is to assess the impact of an innovative strategy to prevent undernutrition and obesity in early childhood in children 0-24 months in Mexico. This study is designed to evaluate the impact of promoting adequate infant an young child feeding practices and the use of SQ-LNS (Small Quantity Lipid-Based Nutrient Supplements) on the nutritional status of infants and young children. The study will be conducted in peri-urban areas of Tepic, Nayarit in Mexico in conjunction with the Hospital Infantil de México Federico Gómez and the Nayarit Secretariat of Health.

DETAILED DESCRIPTION:
SPOON Mexico is an innovative strategy to prevent undernutrition and obesity in children aged 0-24 months living in marginalized areas of Tepic City, Nayarit. The SPOON program aims to improve infant and young children feeding practices, including exclusive breastfeeding, and promote the use of home-fortification with peanut-based SQ-LNS (small quantity lipid-based nutrient supplements) through a novel behavior change strategy.

The study will recruit children between 0 and 6 months of age as well as pregnant women in the third trimester. Mothers or caregivers of eligible children will be invited to participate and a consent form obtain. Participation will start at 0-6 months and the intervention will last until children are up to 24 months. Participants will be randomly assigned at the household level to one of two groups: a control group and a treatment group. Participants in the control group will receive the standard services provided by their local health clinics according to the national protocol. Participants in Treatment Group 1 will receive SQ-LNS supplement from 6-24 months and an innovative behavioral change strategy designed using ethnographic and marketing methods to promote adequate infant and young child feeding practices and the use of SQ-LNS. The strategy will be delivered to mothers or caregivers through individual home-visits and group sessions.

A sample size of 600 children per group has been calculated to detect a minimum effect size of 0.18 with 95% level of significance and a 80% power. Additionally, a 20% attrition has been included in the sample size calculation.

Main outcomes include infant and young child feeding practices, height, weight, hemoglobin, prevalence of anemia, prevalence of stunting, prevalence of obesity, and weight gain rate. A baseline and final survey will be conducted to collect data for these variables, as well as sociodemographic information. Impact estimation will be done comparing the average results and the distribution of indicators between the treatment and control group. Differences of simple means and regression models including co-variables of the child's age and sex, and characteristics of the primary caregiver and household will be estimated. In addition to potential changes in indicator averages, changes in the distribution of variables will be explored under the hypothesis that the intervention might not only improve average value for a given indicator, but compress the distribution over a range of values closer to an optimal range. Changes to distributions will be checked by applying the Kolmogorov-Smirnov test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester and children up to 6 months of age at the moment of recruitment (or children with a maximum age of 6 months at the beginning of the first visit of the program)
* Children with no chronic diseases or congenital malformations
* Resident population from Tepic and the adjacent areas of Xalisco, Lomas Verdes, and Cerro Blanco
* The residents have no plans to move away from Tepic in the following 24 months

Exclusion Criteria:

* Population belonging to the PROSPERA program
* Children with chronic diseases or congenital malformations
* Children with severe acute malnutrition
* Planning on moving far from the intervention area in the next 24 months

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Infant and young child feeding practices at 6 months | Measured at 6 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices at 9 months | Measured at 9 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices at 12 months | Measured at 12 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices 15 months | Measured 15 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices at 18 months | Measured at 18 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices at 21 months | Measured at 21 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Infant and young child feeding practices at 24 months | Measured at 24 months of age
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Height at 6 months | Measured at 6 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 9 months | Measured at 9 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 12 months | Measured at 12 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 15 months | Measured at 15 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 18 months | Measured at 18 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 21 months | Measured at 21 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Height at 24 months | Measured at 24 months of age
  Height-for-age z score obtained by measuring the height of participant children using a fixed infantometer
Weight gain rate at 6 months | Constructed from weight measurements at 6 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 9 months | Constructed from weight measurements at 9 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 12 months | Constructed from weight measurements at 12 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 15 months | Constructed from weight measurements at 15 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 18 months | Constructed from weight measurements at 18 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 21 months | Constructed from weight measurements at 21 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Weight gain rate at 24 months | Constructed from weight measurements at 24 months of age
  Rate of weight gain from 0-24 months of age obtained by measuring the weight of participant children using a fixed electronic scale
Hemoglobin at 6 months | Measured at 6 months of age
  Measurement of hemoglobin concentration in blood using blood biometry
Hemoglobin at 12 months | Measured at 12 months of age
  Measurement of hemoglobin concentration in blood using blood biometry
Hemoglobin at 18 months | Measured at 18 months of age
  Measurement of hemoglobin concentration in blood using blood biometry
Hemoglobin at 24 months | Measured at 24 months of age
  Measurement of hemoglobin concentration in blood using blood biometry
Prevalence of obesity in children at 6 months | Measured at 6 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 9 months | Measured at 9 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 12 months | Measured at 12 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 15 months | Measured at 15 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 18 months | Measured at 18 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 21 months | Measured at 21 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of obesity in children at 24 months | Measured at 24 months of age
  Population estimation of obesity using Body Mass Index (BMI)
Prevalence of stunting at 6 months | Measured at 6 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 9 months | Measured at 9 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 12 months | Measured at 12 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 15 months | Measured at 15 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 18 months | Measured at 18 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 21 months | Measured at 21 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of stunting at 24 months | Measured at 24 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of anemia at 6 months | Measured at 6 months of age
  Population estimation of anemia using hemoglobin concentration in blood
Prevalence of anemia at 12 months | Measured at 12 months of age
  Population estimation of anemia using hemoglobin concentration in blood
Prevalence of anemia at 18 months | Measured at 18 months of age
  Population estimation of anemia using hemoglobin concentration in blood
Prevalence of anemia at 24 months | Measured at 24 months of age
  Population estimation of anemia using hemoglobin concentration in blood

SECONDARY OUTCOMES:
Adherence to Nutritional Supplement Regime | Measured every month from 6 months of age until 24 months of age
  Consumption of the nutritional supplement measured as the number of packets consumed in one month
Exclusive Breastfeeding | Measured 24 months after the start of the intervention
  Measured as an indicator of exclusive breastfeeding, self-reported by the mother of a child

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Martinez, Study Director — Inter-American Development Bank
Locations (1):
- SPOON Mexico, Tepic, Nayarit, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual data will be shared among participating research institutions and made public 2 years after finalizing the study